CLINICAL TRIAL: NCT06700798
Title: A Randomized, Open-Label Phase II Clinical Study of Orelabrutinib Combined With Rituximab Versus R-CVP in the Treatment of Newly Diagnosed Marginal Zone Lymphoma (MZL).
Brief Title: Orelabrutinib Combined With Rituximab Versus R-CVP in the Untreated MZL： A Randomized, Open Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fei Li (Other)
Responsible Party: Sponsor-Investigator, Fei Li, Chief physician, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORRIS
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Marginal Zone Lymphoma(MZL)
Keywords: Orelabrutinib combined with Rituximab versus R-CVP
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; Rituximab; Cyclophosphamide; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OR-R (Experimental): Orelabrutinib 150mg, oral, once daily, Days 1-28, with a cycle of 4 weeks; Cycles 1-24； Rituximab: 375mg/m^2, intravenous, Day 1, with a cycle of 4 weeks; Cycles 1-6
  Interventions: Drug: Orelabrutinib; Drug: rituximab
- R-CVP (Active Comparator): Rituximab: 375mg/m^2, intravenous, Day 1, with a cycle of 3 weeks; Cycles 1-8； Cyclophosphamide: 750mg/m^2, intravenous, Day 1, with a cycle of 3 weeks;Cycles 1-8； Vincristine: 1.4mg/m^2 (maximum 2mg), intravenous, Day 1, with a cycle of 3 weeks;Cycles 1-8； Prednisone: 60mg/m^2, oral, Days 1-5, with a cycle of 3 weeks，Cycles 1-8
  Subsequently, maintenance with rituximab monotherapy until two years from the start of treatment or until toxicity intolerable.
  Interventions: Drug: rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone tablet

INTERVENTIONS:
Drug: Orelabrutinib — 150mg po
  Other Names: ICP-022
  Arms: OR-R
Drug: rituximab — 375mg/m^2, intravenous
Drug: Cyclophosphamide — 750mg/m^2
  Arms: R-CVP
Drug: Vincristine — 1.4mg/m^2
  Arms: R-CVP
Drug: Prednisone tablet — 60mg/m^2
  Arms: R-CVP

SUMMARY:
This study is a randomized, open-label, multicenter, prospective clinical trial aimed at evaluating the efficacy and safety of orelabrutinib combined with rituximab for the previously untreat MZL

DETAILED DESCRIPTION:
For patients with advanced-stage MZL who require treatment, immunochemotherapy is the standard therapy, including regimens such as BR, R-CHOP, R-CVP, etc. The second-generation BTK inhibitor, orelabrutinib, has shown promising efficacy in relapsed/refractory MZL, suggesting that a chemofree regimen combining orelabrutinib with rituximab could also achieve good clinical outcomes in first-line treatment of MZL. However, there is still a lack of prospective studies to confirm this. This study plans to compare the efficacy and safety of orelabrutinib combined with rituximab followed by maintenance therapy with orelabrutinib to the R-CVP regimen.

ELIGIBILITY:
Inclusion Criteria:

1.Age ≥18 years； 2.ECOG performance status level 0~2； 3.Life expectancy of at least 12 weeks; 4.Confirmed CD20-positive marginal zone lymphoma according to the WHO 2008 lymphoma classification criteria, including splenic MZL, nodal MZL, and extranodal MZL subtypes; 5.Measurable lesions detected by enhanced computed tomography (CT) or magnetic resonance imaging (MRI); 6.Indication for treatment according to NCCN guidelines and no prior systemic treatment for MZL; 7.Normal function of major organs; 8.Women of childbearing age must have taken reliable contraceptive measures or undergone a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and must be willing to use appropriate contraceptive methods during the trial period and for 8 weeks after the last administration of the trial medication. For men, they must agree to use appropriate contraceptive methods during the trial period and for 8 weeks after the last administration of the trial medication or have undergone surgical sterilization; 9.The subject voluntarily participates in this study, signs the informed consent form, has good compliance, and cooperates with follow-up.

-

Exclusion Criteria:

1. Patients with central nervous system involvement;
2. History or concurrent other untreated malignant tumors, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, and superficial bladder cancer;
3. Patients with the following cardiovascular diseases: Grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval for males ≥450 ms, for females ≥470 ms); Class III to IV heart failure according to NYHA standards, or echocardiography indicating left ventricular ejection fraction (LVEF) <50%;
4. Coagulation abnormalities (INR >1.5 or prothrombin time (PT) >ULN+4 seconds or APTT >1.5 ULN), with a tendency to bleed or undergoing thrombolytic or anticoagulant therapy;
5. Arterial/venous thrombotic events within 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
6. Known hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.);
7. Major surgical procedures or severe traumatic injuries, fractures, or ulcers within 4 weeks prior to enrollment;
8. Factors that significantly affect the absorption of oral medications, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
9. Active infections requiring antimicrobial treatment (e.g., requiring antibacterial, antiviral drugs, excluding chronic hepatitis B antiviral treatment, antifungal treatment);
10. Active hepatitis B (HBV DNA ≥2000 IU/mL or 104 copies/mL) or hepatitis C (hepatitis C antibody positive, and HCV RNA above the lower limit of detection of the analytical method);
11. History of substance abuse and inability to quit or mental disorders;
12. Participation in other anticancer drug clinical trials within 4 weeks prior to enrollment;
13. Received treatment with potent CYP3A4 inhibitors within 7 days prior to enrollment, or received treatment with potent CYP3A4 inducers within 12 days prior to study participation;
14. Pregnant or breastfeeding women; patients of childbearing potential who are unwilling or unable to use effective contraceptive measures;
15. Other situations judged by the investigator that may affect the conduct of the clinical study and the determination of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2027-12-04 (Estimated)

PRIMARY OUTCOMES:
CRR | up to two years
  The proportion of patients who achieve Complete Remission (CR) at the end of the combined antitumor treatment

SECONDARY OUTCOMES:
ORR | up to two years
  ORR is defined as the percentage of participants with partial or complete response
PFS rate at 24month | Two years after the last patient was enrolled.
  the proportion of patients who have not experienced disease progression or death due to any cause within 2 years of receiving the first dose of the study medication.
Safety parameters | up to 3 years
  Type, frequency, and severity of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, professor, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No